CLINICAL TRIAL: NCT01115504
Title: Thiamine Supplementation in Heart Failure Patients Receiving Full Medical Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Mehdi Mousavi, Azad university
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THF
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Last update posted 2010-12-23 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Heart Failure
Keywords: Thiamine; heart failure
MeSH Terms: conditions — Heart Failure | interventions — Thiamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thiamine (Experimental): Thiamine tablets of 300mg are prescribed for 1 months
  Interventions: Drug: Thiamine
- Plascebo (Placebo Comparator): Tablets of 300mg placebo are prescribed for 1 months
  Interventions: Drug: Thiamine

INTERVENTIONS:
Drug: Thiamine — 300 mg daily for 30 days
  Other Names: Thiamine: brand name: Thiamine Hakim

SUMMARY:
The study is performed to consider the effect of thiamine supplementation on symptoms and signs of patients with heart failure and systolic and diastolic function of left ventricle.

DETAILED DESCRIPTION:
The study is performed to consider the effect of thiamine supplementation versus placebo on symptoms and signs of patients with heart failure systolic and diastolic function of left ventricle.

Heart failure patients (left ventricular ejection fraction (LVEF ≤ 40%) are randomized to receive tablets of 300mg or placebo for 1 months in a double-blind fashion. All subjects will be on stable optimal medical therapy according to the present guidelines for at least 3 months before enrolment. At randomization and at study end, echocardiography by a single observer will be performed and assessment of symptoms and signs and quality of life based on self scoring system (from 1 to 7) and objective physical examinations will be done.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients (left ventricular ejection fraction (LVEF ≤ 40%)
* Optimal medical therapy according to the present guidelines for at least 3 months before enrollment.

Exclusion Criteria:

* Decompensated heart failure
* Renal failure
* COPD
* Asthma
* Uncontrolled hypertension
* Bradycardia or tachycardia which needs increase or decrease in medications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Dyspnea score | 30 days
  scores are given by the patients from 1 to 7 to dyspnea and are reevaluted after 30 days of intervention

SECONDARY OUTCOMES:
Edema score | 30 days
  Edema is scored 1 to 7 by a physician and reevaluated 30days later after intervention
Systolic function | 30 days
  ejection fraction, lateral and septal Sm wave (measured by tissue doppler) are evaluetad by echocardiography before and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Mousavi, Cardiologist, Study Chair — Azad university; Said Namazi, MD, Study Director — Azad university
Locations (1):
- Faculty of medicine, Azad university, Shahrood, Semnan Province, Iran